CLINICAL TRIAL: NCT00240617
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Cross-over Study to Determine the Consistency of Response for Trexima* (Sumatriptan 85mg/Naproxen Sodium 500mg) Administered During the Mild Pain Phase for the Acute Treatment of Multiple Migraine Attacks (*Treximet)
Brief Title: Study Of Treximet, Formerly Known as Trexima, In The Acute Treatment Of Multiple Migraine Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRX103635
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Migraine Disorders
Keywords: consistency of response; migraine; satisfaction; early intervention
MeSH Terms: conditions — Migraine Disorders; Personal Satisfaction | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 1 (Active Comparator): Treximet (sumatriptan/naproxen sodium) formerly known as TREXIMA
  Interventions: Drug: sumatriptan succinate/naproxen sodium
- arm 2 (Placebo Comparator): placebo to match
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sumatriptan succinate/naproxen sodium — comparator
  Arms: arm 1
Drug: placebo — placebo to match
  Arms: arm 2

SUMMARY:
The purpose of this study is to determine the consistency of response for Treximet (formerly known as Trexima) when treating four acute migraine attacks at the mild pain phase and within 1 hour of onset of head pain.

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of physician diagnosed migraine and typically experiences 2-6 migraine attacks per month.
* Typically experiences moderate to severe migraine pain preceded by a mild pain phase.
* Differentiate between mild migraine pain and other headache types.
* Women of childbearing potential must be on adequate contraception.

Exclusion Criteria:

* Pregnant and/or nursing mother.
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Basilar or Hemiplegic migraine.
* History of stroke or transient ischemic attacks (TIA).
* History of epilepsy or treated with anti-epileptics within past 5 years.
* Impaired hepatic or renal function.
* History of gastrointestinal bleeding or ulceration.
* Allergy or hypersensitivity to Aspirin or any other NSAID.
* Allergy or hypersensitivity to triptans.
* Participated in an investigational drug trial in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Score on a 4 pt migraine pain scale for multiple migraine attacks | 2 to 24 hours

SECONDARY OUTCOMES:
Within patient consistency of response, freedom from all migraine pain and symptoms, satisfaction, presence or absence of neck pain/discomfort, sinus pain/pressure, recurrence of head pain, safety and tolerability | 2 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (51):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Avon, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, South Daytona, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Moorestown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valley Stream, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Concinnati, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Salem, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Torgovnick J, Sethi NK, Arsura E. Consistency of response to sumatriptan/naproxen sodium in a placebo-controlled cross-over study. Cephalalgia. 2010 Oct;30(10):1277; author reply 1277-9. doi: 10.1177/0333102409352810. Epub 2010 May 13. No abstract available. PMID 20855373
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TRX103635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register